CLINICAL TRIAL: NCT05821907
Title: Development of the Sexual Health Literacy Scale
Brief Title: Sexual Health Literacy Scale
Acronym: SHLS
Status: Completed | Type: Observational
Sponsor: Nurdan Demirci (Other)
Responsible Party: Sponsor-Investigator, Nurdan Demirci, Prof, Marmara University
Organization: Marmara University (Other)
Other Study IDs: 2023.shls.olmezyalazi
Record Dates: First submitted 2023-04-05; First posted 2023-04-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Sexual Behavior; Literacy; Sexuality
MeSH Terms: conditions — Sexual Behavior; Literacy; Sexuality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: data collection group — The scale development process generally consists of three stages as item production, theoretical analysis and psychometric analysis. The researcher provides theoretical support to the item pool during item production. In the theoretical analysis stage, the content validity of the new scale is evaluated and the first item pool is ensured to reflect the desired structure. In the final stage of the psychometric analysis, the researcher evaluates whether the new scale establishes validity and reliability.

SUMMARY:
According to the World Health Organization, sexual health is a state of well-being related to sexuality as a whole, not just the absence of disease or dysfunction or disability. sexual health; It requires a positive and respectful attitude, free from sexual coercion and discrimination, free of violence, enjoyable and safe experiences. It obliges the respect, protection and fulfillment of the sexual rights of every individual. sexual health; includes a safe and respectful framework free from violence and discrimination; it covers not only the reproductive period, but every age period; different sexual identities and forms of sexual expression, as well as livable and critical gender values, roles, expectations and power dynamics. Insufficient information, difficult access to health services and lack of a guiding structure; It negatively affects young individuals' ability to take responsible decisions with good knowledge about sexuality during their sexual development. Information is obtained from channels where erroneous and incorrect information transfer is intense, and the ways of accessing this information play an important role in the spread of sexual myths in society. Based on all these reasons; This study aimed to develop the Sexual Health Literacy Scale.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 18 who are willing to participate in the study, without psychiatric illness,
* No physical or mental disability
* Able to speak and understand Turkish.

Exclusion Criteria:

* Not willing to participate in the study, with psychiatric illness,
* Physically and mentally handicapped
* 18 years and under,
* Does not speak Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is very difficult to determine what kind of universe individuals over the age of 18 create and to reach the representative group even if it is determined. For this reason, rather than the criterion of representing the universe, it was based on creating a heterogeneous sample group by considering various age groups in a "fit for purpose" way. In this direction, the "snowball sampling" technique, which is one of the non-random sampling types, was preferred. Snowball sampling is a sampling method used in cases where it is difficult to reach the desired population and sample, including quantitative research, especially qualitative research, and the desired sampling frame does not include a large number of sample individuals.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
scale development | 3 month
  The data will be collected with the online data collection tool created by the researchers through the software called google forms. During data collection, the e-mail address of the researchers will be indicated on the form so that the questions of the participants can be answered by the researchers. You will be informed that filling out the data collection form will take an average of 10 minutes for each participant.
  In addition, in order to evaluate the test-retest reliability of the scale, data collection tools will be sent to at least 30 randomly selected individuals from the sample two weeks after the first data collection.
test-retest reliability of the scale | Retest( later 2 weeks)
  In order to evaluate the test-retest reliability of the scale, data collection tools will be sent to at least 30 randomly selected individuals from the sample two weeks after the first data collection. Therefore, after the pre-application, the scale will be applied to 400 people within the scope of the calculated sample, and then, two weeks later, at least 50 people will be re-applied from the individuals to whom the same scale was applied.

CONTACTS AND LOCATIONS:
Overall Officials: Rüveyda Ölmez Yalazı, PhDc, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No